CLINICAL TRIAL: NCT02340260
Title: Effects of Time Efficient Low-volume Interval Exercise on Cardiometabolic Risk Factors in Individuals With Type 2 Diabetes
Brief Title: Time Efficient Exercise in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/801
Record Dates: First submitted 2015-01-07; First posted 2015-01-16 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Exercise; Risk factors; Exercise therapy; Hemoglobin A, Glycosylated
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High intensity interval training (Other): High intensity interval training starts with warming up for 3 minutes at 70 % of maximum heart rate before treadmill training 10x1-minute intervals at 90 % of HRmax, with 75 seconds of active recovery at 70 % of HRmax between each interval. Exercise is completed with a three minute cool down. All training sessions are supervised by an exercise physiologist. Treadmill inclination and/or speed will be adjusted to make sure prescribed intensity is met throughout the intervention.
  Interventions: Behavioral: High intensity interval training
- Sprint interval training (Other): Sprint interval training starts with warming up for 3 minutes at 70 % of maximum heart rate before treadmill training 2x20 seconds of maximum intensity intervals, with 3 minutes and 20 seconds of active recovery at 70 % of HRmax between each interval, followed by 3 minutes cooling down at the same intensity. All training sessions are supervised by an exercise physiologist. Treadmill inclination and/or speed will be adjusted to make sure prescribed intensity is met throughout the intervention.
  Interventions: Behavioral: Sprint interval training

INTERVENTIONS:
Behavioral: High intensity interval training — High intensity exercise during 12 weeks with three weekly training sessions
  Arms: High intensity interval training
Behavioral: Sprint interval training — Sprint interval exercise during 12 weeks with three weekly training sessions
  Arms: Sprint interval training

SUMMARY:
Exercise is considered a cornerstone in the prevention and treatment of type 2 diabetes, but few patients exercise according to guidelines. In this study the effect of two time efficient high intensity exercise protocols on glycemic control and other cardiometabolic risk factors are investigated in patients with type 2 diabetes.The investigators assume that glycemic control is improved more by low-volume high intensity interval training than by extremely low-volume sprint interval training.

DETAILED DESCRIPTION:
The world prevalence of diabetes mellitus for 2010 is estimated to 6.4 % of the adult population, and an increase up to 7.7 % is expected before 2030. 90-95 % individuals with diabetes have type 2 diabetes (T2D).

The complications of T2D lead to substantially increased risk of hypertension, cardiovascular disease (CVD) and the development of heart failure. CVD is the most common cause of death in European adults with diabetes, and the risk of developing CVD is double of that observed in individuals without diabetes. Lowering HbA1c in type 2 diabetes decreases the absolute risk of developing CVD by 5-17 %, as well as decreasing all-cause mortality by 6-15 %.

Individuals with T2D are recommended to exercise moderately or vigorously for at least 150 minutes per week. However, the majority of adults fail to meet the guidelines for even the minimum amount of physical activity, and lack of time is often cited as the main reason.

This research group has previously shown that 4x4 minute high intensity aerobic interval training (AIT) yields significantly greater response on HbA1c, BMI and diastolic dysfunction in patients with T2D with duration <10years in contrast to present recommendations. AIT reduces cardiovascular risk factors more than moderate continuous training in patients with heart failure and metabolic syndrome. In metabolic syndrome, AIT is superior in enhancing endothelial function, insulin signaling in fat and skeletal muscle and in reducing blood glucose. This shows that AIT is a time-efficient and highly effective form of exercise for both patients with T2D and other patient groups.

Recently, even lower training volumes than made use of in the projects presented above, have shown indications of improving glycaemic control in T2D. Only two weeks with a total of six sessions of high intensity training reduces blood glucose significantly in individuals with T2D. Even shorter intervals of all-out activity (2-7 bouts of 20-30 seconds of supramaximal ergometer cycling) was shown to improve both aerobic capacity and a number of metabolic and cardiovascular risk factors after few weeks of training.

However, low-volume high-intensity exercise studies are limited for T2D. The present study aims to compare the effect of two time saving, high intensity exercise protocols on cardiovascular risk factors in patients with type 2 diabetes. The investigators assume that glycemic control is improved more by low-volume high intensity interval training than by extremely low-volume sprint interval training.

ELIGIBILITY:
Inclusion Criteria:

* age 20-65 years
* diagnosed with type 2 diabetes within the past 10 years
* no use of insulin.

Exclusion Criteria:

* known cardiovascular disease- or lung disease, coronary artery disease
* untreated hypertension of ≥140/90 mmHg
* orthopaedic or neurological restrictions
* severe obesity (BMI ≥35)
* pregnancy
* unability to exercise
* drug- or alcohol abuse
* reluctance to sign the consent form
* more reported physical active than recommended in current exercise guidelines

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbA1c) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toril A Nagelhus Hernes, prof, Study Director — Department Circulation and Medical Imaging, NTNU
Locations (1):
- Department Circulation and Medical Imaging, NTNU, Trondheim, Norway

REFERENCES:
- [Result] Revdal A, Hollekim-Strand SM, Ingul CB. Can Time Efficient Exercise Improve Cardiometabolic Risk Factors in Type 2 Diabetes? A Pilot Study. J Sports Sci Med. 2016 May 23;15(2):308-13. eCollection 2016 Jun. PMID 27274669